CLINICAL TRIAL: NCT05773508
Title: Impact of Video Regulation Associated With an Emergency Kit on Night Hospitalizations of the Residents of Nursing Homes in the Emergency Medical Dispatch Center.
Brief Title: Impact of Video Regulation Associated With an Emergency Kit on Night Hospitalizations of the Residents of Nursing Homes.
Acronym: VisioR-EHPAD
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University Hospital, Angers (Other Government)
Responsible Party: Sponsor
Other Study IDs: 2022-120
Record Dates: First submitted 2023-03-03; First posted 2023-03-17 (Actual); Last update posted 2023-03-17 (Actual); Status verified 2023-03

CONDITIONS: Emergencies; Old Age; Debility; Nursing Caries
Keywords: emergency; nursing home; geriatric; telemedicine
MeSH Terms: conditions — Emergencies; Frailty

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Group with video-regulation and using of the emergency kit: Use of video regulation and/or emergency kit → addressing modified by the use of one or the other
  Interventions: Device: Video regulation and emergency kit
- Group without video-regulation and using of the emergency kit: no video-regulation and no use of the emergency kit → addressing patients according to the standard of care

INTERVENTIONS:
Device: Video regulation and emergency kit — Video regulation and emergency kit
  Groups: Group with video-regulation and using of the emergency kit

SUMMARY:
The aim is to evaluate the effectiveness of the device (emergency kit and video-medical control in emergency call centers) in reducing deep night hospitalizations of elderly people living in retirement homes.

DETAILED DESCRIPTION:
Approximately 500,000 elderly people live in a nursing homes in France (1). Few studies concern these subjects: 2% of international research studies (1). Among the subjects hospitalised in the emergency department, those from a nursing home represent a significant proportion of the population, with a proportion of 9 to 37% (2). These are mainly elderly patients who are dependent in the acts of daily life, polypathological and with multiple medications (1,2) and for whom any aggression can lead to hospitalisation, a source of physical and psychological destabilisation (3).

Unplanned hospitalisations are frequent: one resident in ten has been hospitalised in the last three months, and up to five in ten over a full year. Ninety-five percent of the reasons for hospitalisation include cardiac decompensation, the consequences of falls, respiratory disorders, confusion, febrile or non-febrile infections, particularly dermatological, dehydration and gastrointestinal disorders, particularly diarrhoea (4).

These hospitalisations are considered to be avoidable in 7 to 67% of cases, depending on the authors (2). This seems to be explained in particular by the lack of availability of doctors or paramedics to identify or carry out the appropriate technical care or simple complementary examinations (5). During the night, the only staff present in these facilities are often orderlies who are less experienced in assessing emergencies. In a recent study, however, they were the ones who influenced the alert and decided to hospitalise in 40% of cases (6).

The value of specific channels for nursing home patients in reducing avoidable hospitalisations has been highlighted, by favouring short non-emergency channels, particularly for complementary examinations and technical care (7).

The possibility of having a rapid medical assessment on-site, a biological analysis within three hours or the implementation of intravenous hydration would avoid the systematic passage of patients residing in nursing homes through the emergency department. The value of advance directives notifying the non-resuscitation situations desired by the patient would make it possible to further reduce this figure (4).

Inappropriate hospitalisations must therefore be avoided by improving decision-making procedures (8).

The use of video regulation has become more widespread since the SARS-CoV-2 pandemic, allowing continuity of care while minimising the risk of virus transmission. Numerous advantages have emerged from this rapidly developing technology, in particular the possibility of remotely monitoring the progress of the most stable patients, while limiting their movements, and keeping the possibility of calling them in person if necessary. (9) However, the technology of video consultation requires an upgrade in the use of the computer tool by both patients and nursing staff (nurses, doctors). Telephone consultations may be preferred for ease of use, especially for elderly patients, as they will offer less information and more uncertain diagnoses than video consultation (10,11).

A pilot study has shown that video regulation in Emergency Dispatch Center (SAMU C15 in France) is a tool that improves the decision of the regulating doctor in almost 50% of cases, particularly in the case of traumatology (12).

In Maine-et-Loire, emergency kits have been in place since the end of 2022, allowing the prescription of emergency drugs by non-medical staff via video-regulation with the emergency doctor. The aim is to be able to deliver treatments during the night, so that the nursing home doctor can assess the patient's condition in the morning. The emergency kit was developed in collaboration with the EHPAD coordinating doctors, the Emergency Dispatch Center of Angers and the geriatric doctors of the University Hospital of Angers.

The objective of this research is to evaluate this new device. It will compare the rate of night hospitalisation of patients residing in nursing home according to the use or not of visio-regulation coupled with the emergency kit by the Emergency physician working in the Emergency Dispatch Center. At the start of the study, not all the nursing home in the department will be equipped with an emergency kit. We will therefore compare the calls to the Emergency Dispatch Center of the nursing homes with the emergency kit and the use of visio-regulation with the calls from nursing homes that do not yet have this device.

ELIGIBILITY:
Inclusion Criteria:

* Patients residing in a medicalized nursing home equipped with a video-regulation kit (smartphone and emergency kit)
* Nightly call from a paramedical staff to the emergency dispatch center for diagnosis / care / referral to the emergency room between 10 pm and 7 am

Exclusion Criteria:

- Call between 7am and 10pm

Min Age: 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Study Population: All patients for whom nursing home carers called the emergency call centre between 10pm and 7am.
Sampling Method: Probability Sample
Enrollment: 350 (Estimated)
Dates: Start 2023-03-06 (Actual); Primary Completion 2025-03-06 (Estimated); Study Completion 2025-06-06 (Estimated)

PRIMARY OUTCOMES:
Rate of nocturnal hospitalizations | 24 hours
  Evaluating the impact of video-regulation on the rate of nocturnal hospitalizations of patients in a nursing home.

CONTACTS AND LOCATIONS:
Locations (1):
- CHU Angers, Angers, France